CLINICAL TRIAL: NCT05965765
Title: Investigation of the Relationship Between Knee Joint Position Sense and Balance, Function and Reaction Time After Total Knee Arthroplasty
Brief Title: Effection of Total Knee Arthroplasty on Knee Joint
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Principal Investigator, Ayşe Nihal Yurttaş, Research Asistant,Physiotherapist, KTO Karatay University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: E-41901325-200-57879
Record Dates: First submitted 2023-07-20; First posted 2023-07-28 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Total Knee Arthroplasty
Keywords: Arthroplasty; Equilibrium; Knee; Knee joint; Knee prosthesis; Recovery of function; Osteoarthritis; Osteoarthritis-knee; Proprioception; Reaction time
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Total Knee Arthroplasty (Experimental): Individuals who have previously undergone Unilateral total knee arthroplasty
  Interventions: Diagnostic Test: Total knee arthroplasty
- Osteoarthritis without surgery (Experimental): According to Kellgren-Lawrence, individuals diagnosed with osteoarthritis between II and IV
  Interventions: Diagnostic Test: osteoarthritis without surgery
- Control Group (Active Comparator): healthy individuals who have not had any knee problems in the last 6 months
  Interventions: Diagnostic Test: control group

INTERVENTIONS:
Diagnostic Test: Total knee arthroplasty — who got total knee arthroplasty because of osteoarthritis
  Arms: Total Knee Arthroplasty
Diagnostic Test: osteoarthritis without surgery — who has osteoarthritis and didn't get any surgery
  Arms: Osteoarthritis without surgery
Diagnostic Test: control group — healthy people
  Arms: Control Group

SUMMARY:
The aim of this study is to evaluate the joint position sense of individuals diagnosed with knee osteoarthritis and who have undergone unilateral total knee arthroplasty surgery, and to examine the effect of joint position sense on parameters related to balance, physical performance, reaction time, kinesiophobia, pain and stiffness.

Answered the question of the relationship between knee joint position sense, balance, physical performance, reaction time, kinesiophobia levels, pain, stiffness and function in individuals who have undergone knee arthroplasty.

Answered the question of the relationship between knee joint position sense, balance, physical performance, reaction time, kinesiophobia levels, pain, stiffness and function in individuals diagnosed with knee OA who have not undergone surgery.

Answered the question of whether there is a difference between the knee joint position sense values, balance, physical performance, reaction time, kinesiophobia levels, pain, stiffness and function of individuals who have undergone Knee Arthroplasty, individuals diagnosed with Knee OA and healthy individuals.

DETAILED DESCRIPTION:
The aim of this study; To evaluate the joint position sense of individuals who met the inclusion-exclusion criteria of the study by examining the retrospective files of individuals who had previously undergone unilateral total knee arthroplasty surgery due to knee osteoarthritis and whose treatments were completed, and to examine the effect of joint position sense on parameters related to balance, physical performance, reaction time, kinesiophobia, pain and stiffness.It is thought that it will be useful to understand the relationship between the individual's balance, reaction time and physical performance parameters by determining the changes in the joint position sense of individuals who have previously undergone unilateral total knee arthroplasty and individuals with knee osteoarthritis. Also, secondarily; it will shed light on the literature about whether all the evaluated parameters are affected only by the presence of the disease or because of surgery.

ELIGIBILITY:
Inclusion Criteria:

* FOR THE GROUP WITH KNEE ARTROPLASTY SURGERY:

  * Be over the age of 40
  * Having previously undergone unilateral total knee arthroplasty and at least 3 months have passed since
  * Volunteer
* FOR GROUP WITH KNEE OSTEOARTHRITIS:

  * Be over the age of 40
  * Being diagnosed with OA clinically and radiologically (Kellgren-Lawrence II-IV)
  * Not having been exposed to any surgical intervention for the knee Not having received intra-articular injection of the knee in the last 3 months.
  * Volunteer
* FOR THE GROUP OF HEALTHY VOLUNTEERS:

  * Be over the age of 40 Not having knee OA or any knee disease No complaints of knee pain in the last 6 months
  * Volunteer

Exclusion Criteria:

* For all groups:

  * Previous knee surgery (People who have undergone replantation surgery)
  * Individuals who have had lower extremity surgery
  * Pregnancy or lactation Those with lower extremity fractures
  * Those with sensory defects
  * Those diagnosed with malignancy Those with incompletely healed fractures
  * Those with circulatory disorders Those who have infection in the areas around the knee joint
  * Those with metal implants
  * Cancer patients known to be life-threatening
  * People with severe hearing loss or visual impairment
  * People with communication problems Those with uncontrollably high blood pressure People with vestibular problems such as vertigo and balance problems
  * Patients who want to leave the study
  * Patients who cannot continue to work due to developing additional disease

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-04 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Knee Position Sense | baseline
  Knee joint position sense will be evaluated with the mobile application. As the target angle, 15˚, 45˚ and 60˚ knee flexion positions will be determined. For the initial target angle of 15˚ knee flexion, the physiotherapist will passively bring the individual's knee to 15˚ knee flexion and remain in this position for 5 seconds. The individual will be asked to feel and remember this angle, and when he thinks he has come to this angle during the test, he will be asked to say "here" by keeping his knee fixed at that angle. The "estimated target angle" that the person perceives as the "target angle" will be recorded with the phone application. For a target angle, the average of the 3 measurements will be recorded. The deviation angle between the taught target angle and the estimated target angle made by the individual will be calculated.
Balance | baseline
  Berg Balance scale, which has Turkish validity and reliability, will be used in the evaluation of balance. Scale; It consists of 14 parameters that evaluate sitting, standing and standing. These parameters are scored between 0 (unable) and 4 (doing safely). The maximum score is 56. As the score decreases, it will be interpreted as the risk of falling increases and the balance is poor.
Reaction Time | baseline
  Nelson Foot Reaction Test will be used to evaluate the reaction rate. Individuals will be asked to remove their shoes and sit on the stool. The dominant side will be positioned so that the toe is 2.5 cm away from the wall and the heel is 5 cm away from the wall. The observer will hold the 30 cm long wooden ruler on the wall and at the level of the dominant toe of the individual to be evaluated, count backwards from three, one by one and say zero, and leave the ruler. The individual will be asked to hold the falling ruler with the toe and the value on the tip of the foot at the moment he catches the ruler will be recorded in centimeters. The test will be repeated 5 times, and the average of the 3 values other than the lowest and highest values will be recorded in centimeters. The average value obtained will be put into the formula "Reaction Time= √2 x Distance (cm)/980 cm/s2" and the reaction time will be calculated and recorded in seconds.
Physical Performance | baseline
  Timed Up & Go Test (TIGT): This test is frequently used in the evaluation of functional status in individuals with OA and its original name is "Timed Up & Go Test" (TUG). During this test, individuals will be asked to get up from a chair with fixed arms while sitting with their feet in contact with the floor, walk 3 meters, return from the marked place at the end of 3 meters, walk back to the chair and sit on the chair. The duration will be started as soon as the hips of the individuals are out of contact with the chair and stopped when their hips come into contact with the chair after they return, and will be recorded in seconds with a stopwatch.
Kinesiophobia | baseline
  Tampa Kinesiophobia Scale will be used in the evaluation of kinesiophobia. The Tampa Kinesiophobia Scale is a 17-question checklist. It is scored between 1 and 4 points on a Likert scale (1 answer I strongly disagree, 4 answer I strongly agree), 4,8,12,16. The calculation of the questions is done by inverting. The score is determined in the range of 17-68 points, and as the score increases, the fear of movement also increases.
Evaluation of Pain, Function, and Stiffness | baseline
  WOMAC index in order to determine the severity of the clinical findings in the cases and the effects of the current clinical picture on the daily living activities of the patients; osteoarthritis index will be evaluated. WOMAC consists of 3 parts and 24 questions. There are 5 questions in the pain section, 2 questions in the stiffness section, and 17 questions in the physical function section. The total WOMAC value will be obtained by scoring the answers given by the patients as none/mild/moderate/severe/extreme, respectively, between 0 and 4 points. Then, the scores of each section will be collected within itself and the score for that section will be found. High WOMAC values indicate an increase in pain and stiffness and deterioration in physical function. As a result of the study examining the acceptability, reliability, validity and sensitivity of the Turkish version of the WOMAC OA index, it was shown that the Turkish version of the WOMAC index had good content validity.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Nihal YURTTAŞ, master, Principal Investigator — KTO Karatay University
Locations (1):
- KTO Karatay University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yurttas AN, Araci A, Akkoyun Sert O, Ismayilov T. Investigation of knee joint position sensation balance reaction time and function in individuals with knee osteoarthritis and unilateral total knee arthroplasty. J Back Musculoskelet Rehabil. 2025 Oct 27:10538127251387392. doi: 10.1177/10538127251387392. Online ahead of print. PMID 41143951